CLINICAL TRIAL: NCT00744341
Title: A Double-Blind, Placebo-Controlled, Randomized, Multi-Center, Dose-Finding Study of SLV320, a Selective A1 Adenosine Receptor Antagonist, to Evaluate the Effect on Renal Function and Safety in Subjects Hospitalized With Acute Decompensated Heart Failure and Renal Dysfunction (Reno-Defend 1)
Brief Title: Safety and Efficacy Study to Evaluate the Effect of SLV320 on Renal Function in Patients With Worsening Heart Failure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was stopped 29OCT2009 due to strategic drug development considerations
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S320.2.011; 2008-003786-20 (EudraCT Number); 00744341 (Other Grant/Funding Number: NCT/NIH)
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2010-09

CONDITIONS: Acute Decompensated Heart Failure; Renal Dysfunction
Keywords: SLV320; Acute Decompensated Heart Failure (ADHF); chronic heart failure; renal failure; I.V. doses; hospitalization
MeSH Terms: conditions — Renal Insufficiency | interventions — SLV320 compound

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental)
  Interventions: Drug: SLV320
- 2 (Experimental)
  Interventions: Drug: SLV320
- 3 (Experimental)
  Interventions: Drug: SLV320
- 4 (Experimental)
  Interventions: Drug: SLV320
- 5 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SLV320 — 1.25mg i.v. bid
  Arms: 1
Drug: SLV320 — 3.75mg i.v. bid
  Arms: 2
Drug: SLV320 — 7.5mg i.v. bid
  Arms: 3
Drug: SLV320 — 15.0mg i.v. bid
  Arms: 4
Drug: Placebo
  Arms: 5

SUMMARY:
The purpose of this study is to determine the efficacy and safety of IV SLV320 in acute heart failure patients with renal dysfunction.

DETAILED DESCRIPTION:
The purpose of this study is to determine the efficacy and safety of IV SLV320 in acute heart failure patients with renal dysfunction.

ELIGIBILITY:
Inclusion Criteria Renal dysfunction defined as estimated eGFR of 20-80 mL/min; history of systolic or diastolic chronic heart failure of at least 14 days duration for which loop diuretic therapy has been prescribed; clinical evidence for volume overload; BNP ≥ 500 pg/mL or NT-pro-BNP > 2000 pg/mL; hospitalization.

Exclusion Criteria Have low output syndrome, defined as having the need for treatment with I.V. inotropes or vasopressors; Need mechanical ventilation; Have significant stenotic valvular disease (severe aortic or mitral stenosis); Have myocardial infarction or hemodynamically destabilizing significant arrythmias (ventricular tachycardia, bradyarrythmias with slow ventricular rate [<45 bpm] or atrial fibrillation/flutter with a rapid ventricular response of >120 bpm), or electrocardiographic evidence of 2nd degree heart block (Mobitz Type II) or 3rd degree AV-block in the absence of a pacemaker, within 30 days of screening; Have acute myocarditis or hypertrophic obstructive, restrictive, or constrictive cardiomyopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Change in serum creatinine from baseline to Day 14 | Day 14

SECONDARY OUTCOMES:
To compare four SLV320 doses to placebo on the change in the following variables: Dyspnea (Likert Scale and PDA scale), eGFR (MDRD Formula), Subject Global Clinical Assessment Score, Urine Osmolality, Serum Osmolality | Up to Day 3 (Dyspnea); Up to Day 4 (Urine Osmolality); Up to Day 60 (eGFR, Subject Global Clinical Assessment Score, Serum Osmolality)
To compare the effect of four I.V. doses of SLV320 with placebo using the trichotomous endpoint of treatment success, treatment failure, or no change | Up to Day 14
To compare the effect of four I.V. doses of SLV320 with placebo on top of diuretic use | Up to Day 3
To compare the effect of four I.V. doses of SLV320 with placebo using a composite endpoint of all-cause mortality, cardiovascular hospitalization or hospitalization for worsening renal function, in time to event and frequency | Up to Day 180
To determine the pharmacokinetic profile of I.V. SLV320 | Up to Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Bethany, Study Director — Solvay Pharmaceuticals
Locations (105):
- United States (28):
  - S320.2.011 Site # 548, Alameda, California
  - S320.2.011 Site # 566, Banning, California
  - S320.2.011 Site # 551, Inglewood, California
  - S320.2.011 Site # 564, Bridgeport, Connecticut
  - S320.2.011 Site # 505, Hollywood, Florida
  - S320.2.011 Site # 507, Jacksonville, Florida
  - S320.2.011 Site # 532, Riverdale, Georgia
  - S320.2.011 Site # 513, Chicago, Illinois
  - S320.2.011 Site # 561, Indianapolis, Indiana
  - S320.2.011 Site # 526, Owensboro, Kentucky
  - S320.2.011 Site # 504, Natchitoches, Louisiana
  - S320.2.011 Site # 546, Biddeford, Maine
  - S320.2.011 Site # 523, Dearborn, Michigan
  - S320.2.011 Site # 534, Detroit, Michigan
  - S320.2.011 Site # 558, Detroit, Michigan
  - S320.2.011 Site # 508, St Louis, Missouri
  - S320.2.011 Site # 541, Brooklyn, New York
  - S320.2.011 Site # 537, New York, New York
  - S320.2.011 Site # 521, Akron, Ohio
  - S320.2.011 Site # 527, Toledo, Ohio
  - S320.2.011 Site # 528, Philadelphia, Pennsylvania
  - S320.2.011 Site # 510, Colombia, South Carolina
  - S320.2.011 Site # 545, Nashville, Tennessee
  - S320.2.011 Site # 519, Tullahoma, Tennessee
  - S320.2.011 Site # 511, Houston, Texas
  - S320.2.011 Site # 518, San Antonio, Texas
  - S320.2.011 Site # 556, Manitowoc, Wisconsin
  - S320.2.011 Site # 565, Milwaukee, Wisconsin
- S320.2.011 Site # 601, Montreal, Canada
- Chile (3):
  - S320.2.011 Site # 427, Santiago
  - S320.2.011 Site # 433, Viña del Mar
  - S320.2.011 Site # 434, Viña del Mar
- Denmark (6):
  - S320.2.011 Site # 100, Aarhus
  - S320.2.011 Site # 102, Aarhus
  - S320.2.011 Site # 104, Copenhagen
  - S320.2.011 Site # 103, Esbjerg
  - S320.2.011 Site # 106, Frederiksberg
  - S320.2.011 Site # 105, Herning
- France (6):
  - S320.2.011 Site # 125, Dijon
  - S320.2.011 Site # 123, Lille
  - S320.2.011 Site # 121, Paris
  - S320.2.011 Site # 124, Pessac
  - S320.2.011 Site # 126, Pontoise
  - S320.2.011 Site # 128, Toulouse
- Germany (7):
  - S320.2.011 Site # 182, Bad Nauheim
  - S320.2.011 Site # 187, Berlin
  - S320.2.011 Site # 186, Frankfurt
  - S320.2.011 Site # 180, Hanover
  - S320.2.011 Site # 185, Limburg
  - S320.2.011 Site # 190, Mannheim
  - S320.2.011 Site # 188, Weiden
- Italy (6):
  - S320.2.011 Site # 146, Aosta
  - S320.2.011 Site # 145, Cremona
  - S320.2.011 Site # 142, Genova
  - S320.2.011 Site # 149, Milan
  - S320.2.011 Site # 140, Modena
  - S320.2.011 Site # 143, Orbassano
- Poland (16):
  - S320.2.011 Site # 250, Bialystok
  - S320.2.011 Site # 231, Inowrocław
  - S320.2.011 Site # 236, Krakow
  - S320.2.011 Site # 249, Lodz
  - S320.2.011 Site # 243, Oława
  - S320.2.011 Site # 240, Poznan
  - S320.2.011 Site # 247, Przeworsk
  - S320.2.011 Site # 242, Puławy
  - S320.2.011 Site # 251, Płock
  - S320.2.011 Site # 239, Radom
  - S320.2.011 Site # 232, Ruda Śląska
  - S320.2.011 Site # 245, Starogard Gdański
  - S320.2.011 Site # 234, Torun
  - S320.2.011 Site # 248, Torun
  - S320.2.011 Site # 238, Tychy
  - S320.2.011 Site # 233, Wroclaw
- Romania (8):
  - S320.2.011 Site # 265, Baia Mare
  - S320.2.011 Site # 262, Brăila
  - S320.2.011 Site # 260, Bucharest
  - S320.2.011 Site # 263, Bucharest
  - S320.2.011 Site # 267, Bucharest
  - S320.2.011 Site # 264, Suceava
  - S320.2.011 Site # 261, Târgovişte
  - S320.2.011 Site # 266, Timișoara
- Russia (16):
  - S320.2.011 Site # 294, Kazan'
  - S320.2.011 Site # 306, Krasnodar
  - S320.2.011 Site # 290, Moscow
  - S320.2.011 Site # 297, Moscow
  - S320.2.011 Site # 299, Moscow
  - S320.2.011 Site # 301, Moscow
  - S320.2.011 Site # 303, Moscow
  - S320.2.011 Site # 304, Moscow
  - S320.2.011 Site # 305, Moscow
  - S320.2.011 Site # 291, Saint Petersburg
  - S320.2.011 Site # 292, Saint Petersburg
  - S320.2.011 Site # 298, Saint Petersburg
  - S320.2.011 Site # 300, Saint Petersburg
  - S320.2.011 Site # 302, Saint Petersburg
  - S320.2.011 Site # 293, Voronezh
  - S320.2.011 Site # 295, Yaroslavl
- Ukraine (8):
  - S320.2.011 Site # 335, Dnipropetrovsk
  - S320.2.011 Site # 332, Ivano-Frankivsk
  - S320.2.011 Site # 334, Kharkiv
  - S320.2.011 Site # 330, Kyiv
  - S320.2.011 Site # 338, Kyiv
  - S320.2.011 Site # 331, Luhansk
  - S320.2.011 Site # 333, Lutsk
  - S320.2.011 Site # 337, Odesa

REFERENCES:
- [Derived] Pang PS, Mehra M, Maggioni AP, Filippatos G, Middlebrooks J, Turlapaty P, Kazei D, Gheorghiade M; RENO-DEFEND Investigators. Rationale, design, and results from RENO-DEFEND 1: a randomized, dose-finding study of the selective A1 adenosine antagonist SLV320 in patients hospitalized with acute heart failure. Am Heart J. 2011 Jun;161(6):1012-23.e3. doi: 10.1016/j.ahj.2011.03.004. PMID 21641345